CLINICAL TRIAL: NCT01205672
Title: Evaluation of the Molecular Effects of Metformin on the Endometrium in Patients With Endometrial Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0927; NCI-2012-01796 (Registry Identifier: NCI CTRP); CBC 965712 (Other Grant/Funding Number: American Cancer Society IRG)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrium; Gynecologic malignancy; Endometrial adenocarcinoma; Insulin/glucose metabolism; Metformin
MeSH Terms: conditions — Endometrial Neoplasms; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Metformin 850 mg by mouth once daily for at least 7 days, and up to 30 days before surgery.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg by mouth once daily for at least 7 days, and up to 30 days before surgery.

SUMMARY:
The goal of this research study is to learn if metformin can affect endometrial cancer cells in women who do not have diabetes.

Objectives:

Primary Objectives:

1. To determine the molecular effects of metformin and associated physiologic changes in insulin/glucose metabolism on the mTOR (mammalian target of rapamycin) signaling pathway in the endometrium of women with endometrial cancer

Secondary Objectives:

1. To describe the effects of metformin on the histology and proliferation of the endometrium in women with endometrial cancer.
2. To assess the effect of body mass index on the response to treatment with metformin
3. To assess the effect of insulin resistance on the response to treatment with metformin
4. To determine effects of metformin on the serum, urine and DNA biomarkers of women with endometrial cancer.

DETAILED DESCRIPTION:
The Study Drug:

Metformin is designed to treat both diabetes and insulin resistance. Both diabetes and insulin resistance have been linked to endometrial cancer. Although you do not have a diagnosis of diabetes, metformin may still have an affect on your cancer cells.

Study Visit (before taking Metformin):

If you are found eligible to take part in this study, you will have a study visit before you begin taking Metformin. The following tests and procedures will be performed:

* Blood (about 2 tablespoons) and urine will be collected for research to look at different hormone levels.
* If needed, a fasting glucose level will be obtained.
* If you are found not to be eligible your blood, urine, and tissue for research will be discarded.

Study Drug Administration:

You will take metformin, by mouth, 1 time each morning, with breakfast, for at least 7 days and up to 30 days until your scheduled surgery is performed. You will record the dates and times you take metformin on a study drug calendar provided by the study staff. You will not take metformin on the day of your surgery.

Study Tests (on the day of your surgery):

You will bring your study drug calendar to the clinic on the day of your surgery. The following tests and procedures will also be performed:

* Blood (about 2 tablespoons) and urine will be collected for routine tests and to check different hormone levels.
* During surgery, you will have a second endometrial biopsy for biomarker testing.

Length of Study:

You will be off study after your surgical procedure.

This is an investigational study.

Up to 30 women will take part in this study. Up to 25 participants will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed informed consent
2. Patients must have histologically-confirmed endometrial adenocarcinoma, any grade (1, 2, or 3) or a mixed tumor with at least an endometrioid component
3. Patients must be a candidate for surgical staging procedure
4. Patients must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile or they are postmenopausal for greater than 12 months
5. Patients must have a documented non-fasting plasma glucose level of less than or equal to 125 mg/dL. If non-fasting plasma glucose is greater than125 mg/dL, patients must have a fasting plasma glucose level less than or equal to 125 mg/dL
6. Patients must have an adequated renal function of >60cc/min as documented by the Cockcroft Gualt creatinine clearance formula: (140 - age) x (weight Kg) DIVIDED BY Estimated GFR+ 72x serum Creatinine (non-IDMS x 85 (female)
7. Patients must have adequate hepatic function as documented by a serum bilirubin < 2.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor

Exclusion Criteria:

1. Patients with a known history of diabetes mellitus type 1 or 2 or currently taking any hypoglycemic agents
2. Patients who have received metformin or another mTOR inhibitor in the last 2 years
3. Patients with uterine sarcomas
4. Patients who have received prior treatment for endometrial carcinoma with cytotoxic or biologic chemotherapy. Patients who have only received hormonal therapy for endometrial cancer may be included
5. Patients who have undergone definitive surgery including hysterectomy or endometrial ablation
6. Patients who are not surgical candidates
7. Patients with a known hypersensitivity to metformin
8. Patients with metabolic acidosis, acute or chronic, including ketoacidosis or increased risk of lactic acidosis
9. Patients who have a history of excessive alcohol use
10. Patients with a history of congestive heart failure requiring pharmacologic treatment
11. Patients with a known history of HIV
12. Patients older than 80 year of age

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-09-16 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-05-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Increase in s6K Expression | 30 days
  Baseline expression of s6K measured using Western blots, which yield ordinal results (e.g. "weak", "moderate", "strong", etc.). After treatment with metformin, expression again observed, and the percent of patients who have an increase in expression will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org